CLINICAL TRIAL: NCT01092598
Title: The Impact of Neurocognition and Symptomatology on Physical Function Among Older Adults With Schizophrenia
Brief Title: Factors Association With Poor Physical Function in Older Adults With Schizophrenia
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: H54355-35547-O1
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Older adults with schizophrenia are a growing segment of the population yet their physical health status is poor. In order to design effective interventions, the contributing factors must be understood. Current data suggest the side effects of psychiatric medications, sociodemographic factors, and health care disparities are a few of the reasons for the poor physical health. There are only limited data on the impact of psychiatric symptomatology and neurocognition on the physical health of this population. These limited data indicate that worse symptomatology and poorer neurocognition may negatively impact physical functioning, a critical component to optimal physical health. The purpose of this pilot study is to begin to fill this knowledge gap by: 1. examining the relationship between neurocognitive function and physical function and 2. Examining the relationship between schizophrenia symptoms and physical function. 3. Examining the relationship between serum Brain Derived Neurotrophic Factor (BDNF) and physical function. Using a descriptive correlational design, 50 older adults (55+) with schizophrenia or schizoaffective disorder will be assessed. Bivariate associations will be used to examine the relationship between key variables including schizophrenia symptoms as measured by the Positive and Negative Syndrome Scale (PANSS), neurocognitive function as measured with the MATRICS Consensus Cognitive Battery (MCCB), Physical Function as measured objectively by the Timed Get Up and Go (TGUG) test and subjectively with the physical component summary subscale of the 12-item short form health survey (SF-12), and serum BDNF. These pilot data will lay the foundation for a future health promoting intervention.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults older than or equal to 55 with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder that pass a capacity to consent test based on comprehension of the consent form.

Exclusion Criteria:

* Non-English speaking,
* Adults younger than 55,
* No diagnosis of schizophrenia of schizoaffective disorder, and/or
* Not passing a capacity to consent test.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English speaking adults older than or equal to 55 with a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder that pass a capacity to consent test based on comprehension of the consent form.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Physical Function | enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF, San Francisco, California, United States